CLINICAL TRIAL: NCT04344990
Title: Comparison Study of Three Different Methods of Postoperative Pain Management After Total Knee Arthroplasty
Brief Title: Postoperative Pain Management After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Georgios Karpetas, Anesthesiologist MD, University Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10037/23.5.2016
Record Dates: First submitted 2017-04-19; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Postoperative Pain; Knee Arthroplasty
Keywords: epidural analgesia; intra-articular infusion analgesia;; femoral nerve block; total knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Group E- Epidural analgesia (Active Comparator): Continuous epidural infusion (control group) with Ropivacaine 0.2% + clonidine 150μg for postoperative pain management right after the end of the procedure. The PCA pump is programmed with continuous infusion (Ropivacaine 0.2% + clonidine 150μg) 2ml/h and bolus dosage 0,5ml per 15min (max dosage 2ml/h). The epidural catheter is placed preoperatively.
  Interventions: Procedure: Epidural analgesia - Group E
- Group F- Femoral blockade (Active Comparator): Continuous femoral nerve blockade infusion with Ropivacaine 0.2% + clonidine 150μg for postoperative pain management right after the end of the procedure.The PCA pump is programmed with continuous infusion (Ropivacaine 0.2% + clonidine 150μg) 2ml/h and bolus dosage 0,5ml per 15min (max dosage 2ml/h). The femoral catheter is placed preoperatively.
  Interventions: Procedure: Femoral blockade - Group F
- Group I- Intraarticular infusion (Active Comparator): Continuous intraarticular infusion with Ropivacaine 0.2% + clonidine 150μg for postoperative pain management right after the end of the procedure.The PCA pump is programmed with continuous infusion (Ropivacaine 0.2% + clonidine 150μg) 2ml/h and bolus dosage 0,5ml per 15min (max dosage 2ml/h). The intraarticular catheter is placed before the closure of the incision.
  Interventions: Procedure: Intraarticular infusion - Group I

INTERVENTIONS:
Procedure: Epidural analgesia - Group E — Postoperative analgesia with continuous epidural infusion (control group) with Ropivacaine 0.2% + clonidine 150μg with PCA pump (2ml/h and bolus dosage 0,5ml per 15min)
  Arms: Group E- Epidural analgesia
Procedure: Femoral blockade - Group F — Postoperative analgesia with continuous femoral nerve blockade infusion with Ropivacaine 0.2% + clonidine 150μg with PCA pump (2ml/h and bolus dosage 0,5ml per 15min) .
  Arms: Group F- Femoral blockade
Procedure: Intraarticular infusion - Group I — Postoperative analgesia with continuous intraarticular infusion with Ropivacaine 0.2% + clonidine 150μg with PCA pump (2ml/h and bolus dosage 0,5ml per 15min)
  Arms: Group I- Intraarticular infusion

SUMMARY:
The study compares three different analgesic techniques in order to determine which one serves as the optimal method for postoperative pain management after Total Knee Arthroplasty in patients suffering from Osteoarthritis

DETAILED DESCRIPTION:
Prospective, randomized, controlled study. Approval of the study from the University Hospital of Patras Ethics Committee. The Total Knee Arthroplasty procedure is performed always from the same team of Orthopedic surgeons who follow the same technique in each patient for the arthroplasty and the placement of the intraarticular catheter as well. The same team of Anesthesiologists (two Anesthesiologists) performs always the same technique for each analgesic method and is responsible for the patients' perioperative condition concerning anesthesia and analgesia.

Preoperatively, one hour prior to the surgery, all patients receive preemptive multimodal analgesia in the following way; 40mg Parecoxib (iv), 1gr Paracetamol (iv), 150mg Pregabalin (po), 8mg Dexamethasone (iv) και 50mg Ranitidine (iv).

All patients receive subarachnoid anesthesia with Ropivacaine 0.75% (7,5mg/ml) in a dosage of 2-3ml titrated according to patient's age and height.

Three groups

1. Continuous epidural infusion (control group) with Ropivacaine 0.2% + clonidine 150μg.
2. Continuous femoral nerve blockade infusion with Ropivacaine 0.2% + clonidine 150μg.
3. Continuous intraarticular infusion with Ropivacaine 0.2% + clonidine 150μg.

All the catheters remain for 48 hours while the infusion rate is 2ml/h + PCA with 0,5ml/15min and lock-out maximum dose 4/h in total volume of 150ml.

Postoperatively all patients also receive; Parecoxib, Paracetamol, Pregabalin, and Ranitidine up to the third postoperative day (doses titrated).

Rescue analgesia: Tramadol Chloride 50-100mg x 2 /24h depending on patient's age and medical history.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for unilateral total knee arthroplasty (TKA) to treat knee osteoarthritis (OA)
2. Fully conversant in the Greek language
3. Written informed consent to participate in the trial

Exclusion Criteria:

1. Age less than 50 years and greater than 85 years.
2. ASA score >III
3. Pregnancy
4. Subarachnoid anesthesia failure
5. Hypersensitivity/ allergy to certain agent used
6. Participation in other research/ study
7. Severe mental disease (schizophrenia, major depression, severe bipolar disorder, substance abuse)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesia | Up to 3 days
  Pain scores, during rest and movement (active and passive) according to NRS (Numeric Rating Scale) right after the end of the surgery and 2, 4, 6, 12, 24, 36, 48, 60 and 72 hours later (postoperatively)

SECONDARY OUTCOMES:
Mobilization | Up to 3 days
  Time of mobilization (standing, walking in room, walking out of room)
LOS | Up to 3 months
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Fotini Fligou, MD, PhD, Study Chair — University of Patras, Department of Anesthesiology and Critical Care Medicine
Locations (1):
- University Hospital of Patras, Pátrai, Achaia, Greece

IPD SHARING:
Plan to Share IPD: No